CLINICAL TRIAL: NCT03867578
Title: Magnetic Resonance Imaging for Detection of Peritoneal Mesothelioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: IRB18-1101
Record Dates: First submitted 2019-03-05; First posted 2019-03-08 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Mesothelioma; Peritoneal Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exploratory Phase - Standard CT Imaging and HR-MRI (Other): The goal is to test several different novel Magnetic Resonance sequences to determine which gives the best visualization of peritoneal disease.
  Interventions: Diagnostic Test: HR-MRI; Diagnostic Test: Standard CT Imaging
- Testing Phase- Conventional and HR-MRI and Ultrasound (Other): Patients will undergo conventional and HR-MRI imaging as well as abdominal ultrasound to define the performance of these methods.
  Interventions: Diagnostic Test: HR-MRI; Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: HR-MRI — The first 5 patients will undergo HR-MRI scans using different sequence parameters. Results in these patients will then be assessed along with standard CT Imaging to determine which sequences appear to best identify peritoneal disease. The optimal HR-MRI sequences will then be used for the next 19 patients in the Testing phase to formally define their performance compared to standard imaging.
Diagnostic Test: Standard CT Imaging — Standard CT scans will be performed for preoperative imaging in all patients.
  Arms: Exploratory Phase - Standard CT Imaging and HR-MRI
Diagnostic Test: Ultrasound — Ultrasound Elastography will be performed using an FDA-Approved diagnostic GE ultrasound scanner
  Arms: Testing Phase- Conventional and HR-MRI and Ultrasound

SUMMARY:
For cancers, such as mesothelioma, that spread to the lining of the stomach, detecting the cancer is very difficult with CT or MRI scans. Researchers at the University of Chicago want to find out if the new experimental MRI and ultrasound imaging techniques do a better job of detecting these cancers. Researchers will use new MRI and ultrasound techniques to see if it can find evidence of cancer that has spread to the lining of the abdomen, and right now these new techniques are only used for research.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Biopsy-proven MPM
3. Surgery for PM planned at UCM within 60 days
4. Able to tolerate CT, MRI, US scans, and surgery
5. Able to provide written informed consent
6. For women of child bearing age, ability and willingness to use appropriate contraceptive methods before imaging and for a period of 365 days thereafter.

Exclusion Criteria:

1. Pregnancy / Breastfeeding
2. Allergy or intolerance to iodinated or gadolinum contrast dyes
3. Contraindications to CT or MRI imaging including chronic kidney disease with GFR <60mL/min/1.73m2
4. Bioimplants unsuitable for MRI imaging (activated by mechanical, electronic, radiofrequency, or magnetic means), such as cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps
5. Permanent tattoos or eyeliner with magnetic dyes
6. Subjects with shrapnel or metal fragments lodged in the body
7. Anxiety, claustrophobia, or any medical condition that would preclude lying still in an MRI scanner for 1-1.5 hours
8. Cardiac, circulatory, or perspiration problems leading to impaired thermoregulation
9. Respiratory or cardiac impairment limiting the ability to lie flat
10. Inability to breath-hold for MRI acquisition
11. Vascular or aneurysm clips or any other surgical implant that is not MRI-compatible
12. Any other ferromagnetic bioimplant that would be damaged by MRI
13. Mental, cognitive, or mental health impairments that preclude the subject from providing informed consent or adhering to the treatment protocol
14. Subjects unable to adhere to the protocol or communicate effectively with researchers
15. Imprisoned subjects
16. Subjects with history of prior CRS/HIPEC or other peritonectomy surgery that might alter characteristics of the peritoneum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Higher Sensitivity for detection using New High Resolution Contrast Enhanced MRI Imaging Sequences compared to standard MRI | 60 Days
  New HR-MRI sequences will demonstrate greater sensitivity than standard MRI for detecting peritoneal metastases.
Higher sensitivity for detection of peritoneal metastatic disease using Ultrasound Elastography compared to standard MRI | 60 Days
  Ultrasound Elastography will demonstrate greater sensitivity than standard MRI for detecting peritoneal metastases.

SECONDARY OUTCOMES:
The performance of diffusion-weighted MRI in detecting peritoneal disease in patients with malignant peritoneal mesothelioma | 60 days
  Use diffusion-weighted MRI in detecting the per-region sensitivity in patients with MPM
Test high-definition small-voxel MRI imaging sequences for detection of peritoneal disease in MPM | 60 days
  To test HR-MRI sequences for detection of peritoneal disease in MPM focusing on the right hemidiaphragmatic and pelvic spaces
Perform Ultrasound Elastography in peritoneal mesothelioma to determine optimal strain ratios | 60 days
  Ultrasound Elastography to determine optimal strain ratios to maximize sensitivity in PM patients
Perform Ultrasound Elastography in peritoneal mesothelioma to determine elasticity scores | 60 days
  Ultrasound Elastography to determine elasticity scores to maximize sensitivity in PM patients

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, MD, Principal Investigator — University of Chicago
Locations (1):
- University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States